CLINICAL TRIAL: NCT00996528
Title: Neighborhood Alcohol & HIV Prevention in South African Townships (Philani)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Mary Jane Rotheram-Borus, Professor, Semel Institute and the Department of Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Federal Identifier # AA017104; I R0I AA017104-01
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Fetal Alcohol Syndrome; HIV; Nutrition Disorders
Keywords: fetal alcohol syndrome; alcohol abuse; HIV; malnutrition; children; mentor mother; behavioral intervention; South Africa; Maternal alcohol use; HIV-related transmission behaviors; low birth weight babies and low-weight children; HIV Seronegativity
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Nutrition Disorders; Alcoholism; Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Philani Intervention Program (Experimental)
  Interventions: Behavioral: Philani Intervention Program
- Standard Care (No Intervention): No intervention during study. Referral to clinic-based health care that is delivered by the province. Offered intervention at end of study, i.e. after 18 months.

INTERVENTIONS:
Behavioral: Philani Intervention Program — Offered to pregnant women / mothers through mentor mothers, i.e. mothers in community who are selected because they are doing well. They are trained to conduct home visits, 2 times a months through pregnancy. After childbirth, visits are spaced depending on the perceived need. If the baby is thriving and mother is coping well with health risks, mentor mother will visit once a month.
  Arms: Philani Intervention Program

SUMMARY:
The purpose of this study is to test a mother-to-mother intervention during pregnancy and after delivery with mothers in South Africa, most of whom are at risk delivering babies with fetal alcohol syndrome, babies that are underweight, or babies that are infected with HIV from an HIV-positive mother. The investigators hypothesize that the intervention will reduce the chance of these three health outcomes occurring in the babies and improve the health of the mother.

DETAILED DESCRIPTION:
There are four intersecting epidemics among pregnant women in South Africa: hazardous alcohol use (30%), HIV (27%), TB (60% of HIV+), and malnutrition (24% of infants). Unless the prevention programs for these epidemics are horizontally integrated, there will never be adequate resources to address these challenges and stigma will dramatically reduce program utilization. Furthermore, while clinics are the typical sites for treating each of these health problems, this proposal will examine a home-visiting prevention program delivered by neighborhood Mentor Mothers (MM) as an alternative to clinic-based interventions to reduce the consequences of hazardous alcohol use, HIV, TB, and poor nutrition. The intervention will encourage mothers to care for their own health, parent well, maintain their mental health, and, if the mother is living with HIV (HIV+ MAR), reduce HIV transmission and/or reduce alcohol use and abuse. The results begin to inform the optimal delivery strategy for next generation of preventive interventions in order to be feasible and sustainable for broad dissemination immediately following an efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman and their children
* Age 18 or older
* Informed consent

Exclusion Criteria:

* Psychosis, neurological damage, inability to communicate with interviewer
* Inability to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1239 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
HIV-related transmission acts | 18 months
  Maternal HIV transmission acts
Baby's health status | 18 months
  Children's behavioral and cognitive adjustment and school achievement
Maternal adherence to HIV-related and general health routines | 18 months
  Maternal alcohol use on the AUDIT
Mental health | 18 months
  Maternal Depression on the Edinburgh Postnatal Depression Scale (EPDS)
Social support | 18 months
  Children's peer relationships at seven and a half years

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane Rotheram-Borus, PhD, Principal Investigator — Department of Psychiatry & Biobehavioral Sciences, Semel Institute, UCLA
Locations (1):
- Philani Child Health and Nutrition Project, Khayelitsha, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data up to the eighth year post birth is being shared with researcher from other institutions.

REFERENCES:
- [Derived] Asarnow LD, Norwood PP, Christodoulou J, Tomlinson M, Rotheram-Borus MJ. The Concurrent and Longitudinal Relationship between Perinatal Sleep Difficulties and Depression in a Large Sample of High-Risk Women in South Africa. Matern Child Health J. 2024 Apr;28(4):700-707. doi: 10.1007/s10995-023-03850-x. Epub 2023 Dec 19. PMID 38110851
- [Derived] Rotheram-Borus MJ, Tomlinson M, Worthman CM, Norwood P, le Roux I, O'Connor MJ. Maternal depression, alcohol use, and transient effects of perinatal paraprofessional home visiting in South Africa: Eight-year follow-up of a cluster randomized controlled trial. Soc Sci Med. 2023 May;324:115853. doi: 10.1016/j.socscimed.2023.115853. Epub 2023 Mar 23. PMID 37001280
- [Derived] Christodoulou J, Rotheram-Borus MJ, Hayati Rezvan P, Comulada WS, Stewart J, Almirol E, Tomlinson M. Where you live matters: Township neighborhood factors important to resilience among south African children from birth to 5 years of age. Prev Med. 2022 Apr;157:106966. doi: 10.1016/j.ypmed.2022.106966. Epub 2022 Jan 20. PMID 35065975
- [Derived] Christodoulou J, Rotheram-Borus MJ, Hayati Rezvan P, Weiss RE, Tomlinson M. Association of early migration with child growth, cognition and behaviour in South Africa. Trop Med Int Health. 2022 Mar;27(3):218-225. doi: 10.1111/tmi.13719. Epub 2022 Jan 23. PMID 34997984
- [Derived] Gordon S, Rotheram-Fuller E, Rezvan P, Stewart J, Christodoulou J, Tomlinson M. Maternal depressed mood and child development over the first five years of life in South Africa. J Affect Disord. 2021 Nov 1;294:346-356. doi: 10.1016/j.jad.2021.07.027. Epub 2021 Jul 16. PMID 34315096
- [Derived] Yonemoto N, Nagai S, Mori R. Schedules for home visits in the early postpartum period. Cochrane Database Syst Rev. 2021 Jul 21;7(7):CD009326. doi: 10.1002/14651858.CD009326.pub4. PMID 34286512
- [Derived] Rotheram-Borus MJ, Christodoulou J, Hayati Rezvan P, Comulada WS, Gordon S, Skeen S, Stewart J, Almirol E, Tomlinson M. Maternal HIV does not affect resiliency among uninfected/HIV exposed South African children from birth to 5 years of age. AIDS. 2019 Jun 1;33 Suppl 1(Suppl 1):S5-S16. doi: 10.1097/QAD.0000000000002176. PMID 31397718
- [Derived] Rotheram-Borus MJ, Arfer KB, Christodoulou J, Comulada WS, Stewart J, Tubert JE, Tomlinson M. The association of maternal alcohol use and paraprofessional home visiting with children's health: A randomized controlled trial. J Consult Clin Psychol. 2019 Jun;87(6):551-562. doi: 10.1037/ccp0000408. PMID 31120274
- [Derived] Tomlinson M, Rotheram-Borus MJ, Harwood J, le Roux IM, O'Connor M, Worthman C. Community health workers can improve child growth of antenatally-depressed, South African mothers: a cluster randomized controlled trial. BMC Psychiatry. 2015 Sep 23;15:225. doi: 10.1186/s12888-015-0606-7. PMID 26400691
- [Derived] Rotheram-Borus MJ, Tomlinson M, le Roux IM, Harwood JM, Comulada S, O'Connor MJ, Weiss RE, Worthman CM. A cluster randomised controlled effectiveness trial evaluating perinatal home visiting among South African mothers/infants. PLoS One. 2014 Oct 23;9(10):e105934. doi: 10.1371/journal.pone.0105934. eCollection 2014. PMID 25340337
- [Derived] le Roux IM, Tomlinson M, Harwood JM, O'Connor MJ, Worthman CM, Mbewu N, Stewart J, Hartley M, Swendeman D, Comulada WS, Weiss RE, Rotheram-Borus MJ. Outcomes of home visits for pregnant mothers and their infants: a cluster randomized controlled trial. AIDS. 2013 Jun 1;27(9):1461-71. doi: 10.1097/QAD.0b013e3283601b53. PMID 23435303